CLINICAL TRIAL: NCT01108263
Title: The Use of INTEGRA™ Flowable Wound Matrix to Manage Diabetic Foot Ulcers in High Risk Populations: A Prospective, Randomized, Controlled Trial
Brief Title: Use of INTEGRA™ Flowable Wound Matrix to Manage Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor Terminated
Sponsor: Georgetown University (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, John Steinberg, DPM, Principle Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-006
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes; Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer | interventions — Collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integra Flowable on wound bed (Active Comparator): INTEGRA™ Flowable is a wound Matrix made of bovine (cow) collagen. It provides a scaffold for cellular and capillary growth. Dosage is dependent on the size of the wound. It will be applied once.
  Interventions: Drug: INTEGRA™ Flowable Matrix (Collagen)
- INTEGRA Flowable on wound & injected subcutaneously (Active Comparator): INTEGRA™ Flowable is a wound Matrix made of bovine (cow) collagen. It provides a scaffold for cellular and capillary growth. Dosage is dependent on the size of the wound. It will be applied once.
  Interventions: Drug: INTEGRA™ Flowable Matrix (Collagen)

INTERVENTIONS:
Drug: INTEGRA™ Flowable Matrix (Collagen) — INTEGRA™ Flowable Wound Matrix is an advanced 3-D porous matrix comprised of granulated cross-linked bovine tendon collagen and glycosaminoglycan. It provides a scaffold for cellular invasion and capillary growth. The collagen and glycosaminoglycan mix is hydrated with saline and applied on the wound bed.
  Other Names: Integra Flowable Wound Matrix

SUMMARY:
* After determining if subjects meet the criteria to be included in the study they will be randomly placed in either Group 1 or 2 and patient will be blinded from randomization group.
* Subjects will walk across a pressure plate to determine different areas of high pressure under the foot. This will be done before the INTEGRA application and at every other follow-up visit.
* Both groups will be debrided and have pictures taken in the OR
* Group 1 will have Integra Flowable Wound Matrix applied onto the wound in the OR and Group 2 will have the Integra Flowable Wound Matrix applied onto the wound and injected subcutaneously in the OR.
* Subjects will be placed in a total contact cast at each visit.

If wound healing occurs prior to 12 weeks, a final assessment visit will be done and the status of the healed ulcer will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subjects with a plantar diabetic foot wound, with or without a previous history of partial foot amputation.
3. Subject has Diabetes Mellitus (type 1 or type 2).
4. University of Texas Classification 1A with a wound area measurement ranging between 0.3-4.0cm².
5. Ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study.

Exclusion Criteria:

1. Subjects < 18 years of age
2. Subject is non-diabetic
3. Subjects who present with wounds of etiology other than diabetes
4. Subject demonstrates increased signs of clinical infection
5. Has active malignant disease of any kind. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
6. University of Texas Classification greater than grade 1A
7. Diabetic plantar foot wounds measuring >4.0cm²
8. Subjects who present with significant vascular or metabolic comorbidity that would preclude wound healing
9. Subjects participating in any other trials in regards to the diabetic foot ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Steinberg, DPM, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integra Flowable on Wound Bed | INTEGRA Flowable on Wound & Injected Subcutaneously
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integra Flowable on Wound Bed | INTEGRA Flowable on Wound & Injected Subcutaneously | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (0.70711) | 47 (4.58258) | 50 (5.24404)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Decrease in Wound Size
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Integra Flowable on Wound Bed | INTEGRA Flowable on Wound & Injected Subcutaneously
Number analyzed (Participants) | 2 | 3
participants | 2 | 2

2. Secondary Outcome: Decreased Peak Plantar Pressures in Both the Static and Dynamic Phases of Gait as Compared to Pre-operative Pressure Values.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Integra Flowable on Wound Bed | INTEGRA Flowable on Wound & Injected Subcutaneously
Number analyzed (Participants) | 2 | 3
participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Integra Flowable on Wound Bed | INTEGRA Flowable on Wound & Injected Subcutaneously
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Integra Flowable on Wound Bed (N=2) | INTEGRA Flowable on Wound & Injected Subcutaneously (N=3)
Wound infection (Skin and subcutaneous tissue disorders) | 0 | 1
Chest pain (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other